CLINICAL TRIAL: NCT05932693
Title: Examine the Effects of Novel E-cigarette Constituents and Determining Appropriate Concentrations Among Adults
Brief Title: Effect of Different E-cigarette Cooling Flavors on Adults' Sensory Experience TCORS 3.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2000035551_a; 2U54DA036151-11 (NIH)
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: E-Cig Use
Keywords: Cooling components; e-cigarette; menthol; WS-23; WS-3
MeSH Terms: conditions — Vaping | interventions — Menthol

STUDY DESIGN:
Intervention Model Description: Participants are exposed to all study conditions (16 e-liquid samples).
Who Masked: Participant, Investigator
Masking Description: Participants will be exposed to e-liquids containing 16 conditions (WS-3 block: 0.05%, 0.1%, 0.5%, 1.0%, 2.0%, WS-23 block: 0.05%, 0.1%, 0.5%, 1.0%, 2.0%, 4.0%, and menthol block: 0.05%, 0.1%, 0.5%, 1.0%, 2.0%) from low concentration to high concentration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- WS-3 (1), no nicotine (Experimental): WS-3 block: 0.05%
  Interventions: Other: E-liquid coolant (WS-3, 0.05%)
- WS-3 (2), no nicotine (Experimental): WS-3 block: 0.1%
  Interventions: Other: E-liquid coolant (WS-3, 0.1%)
- WS-3 (3), no nicotine (Experimental): WS-3 block: 0.5%
  Interventions: Other: E-liquid coolant (WS-3, 0.5%)
- WS-3 (4), no nicotine (Experimental): WS-3 block: 1.0%
  Interventions: Other: E-liquid coolant (WS-3, 1.0%)
- WS-3 (5), no nicotine (Experimental): WS-3 block: 2.0%
  Interventions: Other: E-liquid coolant (WS-3, 2.0%)
- Menthol (1), no nicotine (Experimental): Menthol block: 0.05%
  Interventions: Other: E-liquid coolant (menthol, 0.05%)
- Menthol (2), no nicotine (Experimental): Menthol block: 0.1%
  Interventions: Other: E-liquid coolant (menthol, 0.1%)
- Menthol (3), no nicotine (Experimental): Menthol block: 0.5%
  Interventions: Other: E-liquid coolant (menthol, 0.5%)
- Menthol (4), no nicotine (Experimental): Menthol block: 1.0%
  Interventions: Other: E-liquid coolant (menthol, 1.0%)
- Menthol (5), no nicotine (Experimental): Menthol block: 2.0%
  Interventions: Other: E-liquid coolant (menthol, 2.0%)
- WS-23 (1), no nicotine (Experimental): WS-23 block: 0.05%
  Interventions: Other: E-liquid coolant (WS-23, 0.05%)
- WS-23 (2), no nicotine (Experimental): WS-23 block: 0.1%
  Interventions: Other: E-liquid coolant (WS-23, 0.1%)
- WS-23 (3), no nicotine (Experimental): WS-23 block: 0.5%
  Interventions: Other: E-liquid coolant (WS-23, 0.5%)
- WS-23 (4), no nicotine (Experimental): WS-23 block: 1.0%
  Interventions: Other: E-liquid coolant (WS-23, 1.0%)
- WS-23 (5), no nicotine (Experimental): WS-23 block: 2.0%
  Interventions: Other: E-liquid coolant (WS-23, 2.0%)
- WS-23 (6), no nicotine (Experimental): WS-23 block: 4.0%
  Interventions: Other: E-liquid coolant (WS-23, 4.0%)

INTERVENTIONS:
Other: E-liquid coolant (WS-3, 0.05%) — Adult users of e-cigarette will be exposed to five e-liquid coolants WS-3: 0.05%.
  Other Names: Flavor type
  Arms: WS-3 (1), no nicotine
Other: E-liquid coolant (WS-3, 0.1%) — Adult users of e-cigarette will be exposed to five e-liquid coolants WS-3: 0.1%.
  Other Names: Flavor type
  Arms: WS-3 (2), no nicotine
Other: E-liquid coolant (WS-3, 0.5%) — Adult users of e-cigarette will be exposed to five e-liquid coolants WS-3: 0.5%.
  Other Names: Flavor type
  Arms: WS-3 (3), no nicotine
Other: E-liquid coolant (WS-3, 1.0%) — Adult users of e-cigarette will be exposed to five e-liquid coolants WS-3: 1.0%.
  Other Names: Flavor type
  Arms: WS-3 (4), no nicotine
Other: E-liquid coolant (WS-3, 2.0%) — Adult users of e-cigarette will be exposed to five e-liquid coolants WS-3: 2.0%.
  Other Names: Flavor type
  Arms: WS-3 (5), no nicotine
Other: E-liquid coolant (menthol, 0.05%) — Adult users of e-cigarette will be exposed to five e-liquid coolants menthol: 0.05%.
  Other Names: Flavor type
  Arms: Menthol (1), no nicotine
Other: E-liquid coolant (menthol, 0.1%) — Adult users of e-cigarette will be exposed to five e-liquid coolants menthol: 0.1%.
  Other Names: Flavor type
  Arms: Menthol (2), no nicotine
Other: E-liquid coolant (menthol, 0.5%) — Adult users of e-cigarette will be exposed to five e-liquid coolants menthol: 0.5%.
  Other Names: Flavor type
  Arms: Menthol (3), no nicotine
Other: E-liquid coolant (menthol, 1.0%) — Adult users of e-cigarette will be exposed to five e-liquid coolants menthol: 1.0%.
  Other Names: Flavor type
  Arms: Menthol (4), no nicotine
Other: E-liquid coolant (menthol, 2.0%) — Adult users of e-cigarette will be exposed to five e-liquid coolants menthol: 2.0%.
  Other Names: Flavor type
  Arms: Menthol (5), no nicotine
Other: E-liquid coolant (WS-23, 0.05%) — Adult users of e-cigarette will be exposed to six e-liquid coolants WS-23: 0.05%.
  Other Names: Flavor type
  Arms: WS-23 (1), no nicotine
Other: E-liquid coolant (WS-23, 0.1%) — Adult users of e-cigarette will be exposed to six e-liquid coolants WS-23: 0.1%.
  Other Names: Flavor type
  Arms: WS-23 (2), no nicotine
Other: E-liquid coolant (WS-23, 0.5%) — Adult users of e-cigarette will be exposed to six e-liquid coolants WS-23: 0.5%.
  Other Names: Flavor type
  Arms: WS-23 (3), no nicotine
Other: E-liquid coolant (WS-23, 1.0%) — Adult users of e-cigarette will be exposed to six e-liquid coolants WS-23: 1.0%.
  Other Names: Flavor type
  Arms: WS-23 (4), no nicotine
Other: E-liquid coolant (WS-23, 2.0%) — Adult users of e-cigarette will be exposed to six e-liquid coolants WS-23: 2.0%.
  Other Names: Flavor type
  Arms: WS-23 (5), no nicotine
Other: E-liquid coolant (WS-23, 4.0%) — Adult users of e-cigarette will be exposed to six e-liquid coolants WS-23: 4.0%.
  Other Names: Flavor type
  Arms: WS-23 (6), no nicotine

SUMMARY:
This pilot sensory experiment will examine cooling from comparable concentrations of WS-3 and menthol to determine appropriate concentrations to use in the main study.

DETAILED DESCRIPTION:
This pilot study will establish low and high concentrations of both WS-3 and menthol concentrations to test in the main study. An anticipated 30 adult e-cigarette users will participate in one laboratory session during which participants will be exposed to e-liquids containing five different concentrations of two different cooling flavors without nicotine (10 e-liquids total). Participants will rate "coolness" using the generalized Labeled Magnitude Scale (gLMS). Using averages of participant ratings, we will select a low concentration of each constituent that is rated as more than "barely detectable" but less than "moderate" to ensure that cooling is weak but clearly perceptible. For the high concentration of each constituent, we will select a concentration that on average falls between "strong" and "very strong" to identify a strong cooling sensation while avoiding sensations that would also be uncomfortable.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to read and write
* Used e-cigarettes containing nicotine
* Use e-cigs in past 30 days
* No strong dislike of the menthol flavor
* Urine cotinine ≥200ng/ml
* Willing to abstain from tobacco/nicotine use 2 hrs prior to sessions

Exclusion Criteria:

* Known hypersensitivity to propylene glycol
* Pregnant or lactating females
* Uncontrolled asthma
* Nut/e-liquid flavorant allergy
* Current marijuana (tetrahydrocannabinol) vaping + E-cigarette or vaping use Associated Lung Injury (EVALI) symptoms
* Dislike of menthol flavor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
We may share information about the IPD and study results with other researchers in the future, but the information will be de-identified.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The identifiable information will be kept for 7 years. After that, the data will become anonymous.
Access Criteria: The de-identified data will be made available for research purposes by contacting the PI.

REFERENCES:
- [Background] Lim J, Wood A, Green BG. Derivation and evaluation of a labeled hedonic scale. Chem Senses. 2009 Nov;34(9):739-51. doi: 10.1093/chemse/bjp054. PMID 19833660

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the local community and university settings using flyers, email advertisements, and online postings. Individuals who expressed interest were screened for eligibility and checked during intakes, and those meeting inclusion criteria were scheduled for a single laboratory session. A total of 31 eligible participants were enrolled, and 30 completed the study procedures, 27 were analyzed
Pre-assignment Details: Prior to completion of the lab session, one participant did not attend (due to no-show) and was therefore excluded from the final dataset. A total of 30 participants completed the laboratory procedures and were assigned to the study conditions.
Groups:
- A Single Lab Session With 16 Conditions/Exposures: Participants attended a lab session that included 16 conditions/exposures involving WS-3, WS-23, and menthol. The three types of coolants were presented in randomized blocks, with each block containing increasing concentrations. The specific 16 conditions are listed below:
  WS-3 block (1): 0.05%, no nicotine; WS-3 block (2): 0.1%, no nicotine; WS-3 block (3): 0.5%, no nicotine; WS-3 block (4): 1.0%, no nicotine; WS-3 block (5): 2.0%, no nicotine; Menthol block (1): 0.05%, no nicotine; Menthol block (2): 0.1%, no nicotine; Menthol block (3): 0.5%, no nicotine; Menthol block (4): 1.0%, no nicotine; Menthol block (5): 2.0%, no nicotine; WS-23 block (1): 0.05%, no nicotine; WS-23 block (2): 0.1%, no nicotine; WS-23 block (3): 0.5%, no nicotine; WS-23 block (4): 1.0%, no nicotine; WS-23 block (5): 2.0%, no nicotine; WS-23 block (6): 4.0%, no nicotine
Period: Overall Study
Arm/Group | A Single Lab Session With 16 Conditions/Exposures
Started | 31
WS-3 block (1): 0.05%, no nicotine | 30
WS-3 block (2): 0.1%, no nicotine | 30
WS-3 block (3): 0.5%, no nicotine | 30
WS-3 block (4): 1.0%, no nicotine | 30
WS-3 block (5): 2.0%, no nicotine | 30
Menthol block (1): 0.05%, no nicotine | 30
Menthol block (2): 0.1%, no nicotine | 30
Menthol block (3): 0.5%, no nicotine | 30
Menthol block (4): 1.0%, no nicotine | 30
Menthol block (5): 2.0%, no nicotine | 30
WS-23 block (1): 0.05%, no nicotine | 30
WS-23 block (2): 0.1%, no nicotine | 30
WS-23 block (3): 0.5%, no nicotine | 30
WS-23 block (4): 1.0%, no nicotine | 30
WS-23 block (5): 2.0%, no nicotine | 30
WS-23 block (6): 4.0%, no nicotine | 30
Completed | 30
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the 31 participants who were eligible to attend the lab session.
Arm/Group | A Single Lab Session With 16 Conditions/Exposures
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years old] | 33.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 16
  Non-Hispanic Black | 7
  Non-Hispanic Asian | 4
  Hispanic or Latino | 3
  Others | 1
E-cigarette use frequency [Mean (Standard Deviation); unit: days] — Mean number of days used in past 28 days
  days | 26.0 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Coolness: Score Change in Coolness of Each E-cigarette Condition (16 Conditions in Total)
Description: Difference in overall flavor intensity, coolness, sweetness and harshness/irritation at each e-cigarette condition as measured by the computerized Generalized Labeled Magnitude Scale (gLMS). Participants will self-report their responses using a computer mouse to indicate where on the scale response falls. The Generalized Labeled Magnitude Scales (gLMS) are category ratio scales with seven semantic labels: "no sensation", "barely detectable", "weak", "moderate", "strong", "very strong", and "strongest imaginable", positioned quasi-logarithmically as per empirically determined semantic magnitudes on a 0-100 scale (strongest imaginable at the 100 end).
Time Frame: Following administration of e-cigarette condition 1 (at 10 minutes), then 5 minutes post administration of each e-cigarette condition, up to 85 minutes (condition 16)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- WS-3 (1), 0.05%: WS-3 block: 0.05%, no nicotine
- WS-3 (2), 0.1%: WS-3 block: 0.1%, no nicotine
- WS-3 (3), 0.5%: WS-3 block: 0.5%, no nicotine
- WS-3 (4), 1.0%: WS-3 block: 1.0%, no nicotine
- WS-3 (5), 2.0%: WS-3 block: 2.0%, no nicotine
- Menthol (1), 0.05%: Menthol block: 0.05%, no nicotine
- Menthol (2), 0.1%: Menthol block: 0.1%, no nicotine
- Menthol (3), 0.5%: Menthol block: 0.5%, no nicotine
- Menthol (4), 1.0%: Menthol block: 1.0%, no nicotine
- Menthol (5), 2.0%: Menthol block: 2.0%, no nicotine
- WS-23 (1), 0.05%: WS-23 block: 0.05%, no nicotine
- WS-23 (2), 0.1%: WS-23 block: 0.1%, no nicotine
- WS-23 (3), 0.5%: WS-23 block: 0.5%, no nicotine
- WS-23 (4), 1.0%: WS-23 block: 1.0%, no nicotine
- WS-23 (5), 2.0%: WS-23 block: 2.0%, no nicotine
- WS-23 (6), 4.0%: WS-23 block: 4.0%, no nicotine
Arm/Group | WS-3 (1), 0.05% | WS-3 (2), 0.1% | WS-3 (3), 0.5% | WS-3 (4), 1.0% | WS-3 (5), 2.0% | Menthol (1), 0.05% | Menthol (2), 0.1% | Menthol (3), 0.5% | Menthol (4), 1.0% | Menthol (5), 2.0% | WS-23 (1), 0.05% | WS-23 (2), 0.1% | WS-23 (3), 0.5% | WS-23 (4), 1.0% | WS-23 (5), 2.0% | WS-23 (6), 4.0%
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27 | 27
Scores on a scale | 2.70 (3.47) | 3.35 (5.78) | 5.43 (4.80) | 8.13 (6.15) | 11.61 (13.07) | 3.91 (7.37) | 4.14 (5.43) | 11.18 (11.23) | 12.23 (7.92) | 18.65 (12.54) | 4.52 (6.12) | 3.17 (4.21) | 8.22 (9.20) | 12.57 (11.21) | 17.69 (10.58) | 28.46 (15.37)

ADVERSE EVENTS:
Time Frame: Participants complete an intake assessment and a single laboratory visit, with all assessments completed within approximately 2 weeks of enrollment.
Groups:
- WS-3 Block (1): 0.05%: WS-3 block (1): 0.05%, no nicotine
- WS-3 Block (2): 0.1%: WS-3 block (2): 0.1%, no nicotine
- WS-3 Block (3): 0.5%: WS-3 block (3): 0.5%, no nicotine
- WS-3 Block (4): 1.0%: WS-3 block (4): 1.0%, no nicotine
- WS-3 Block (5): 2.0%: WS-3 block (5): 2.0%, no nicotine
- Menthol Block (1): 0.05%: Menthol block (1): 0.05%, no nicotine
- Menthol Block (2): 0.1%: Menthol block (2): 0.1%, no nicotine
- Menthol Block (3): 0.5%: Menthol block (3): 0.5%, no nicotine
- Menthol Block (4): 1.0%: Menthol block (4): 1.0%, no nicotine
- Menthol Block (5): 2.0%: Menthol block (5): 2.0%, no nicotine
- WS-23 Block (1): 0.05%: WS-23 block (1): 0.05%, no nicotine
- WS-23 Block (2): 0.1%: WS-23 block (2): 0.1%, no nicotine
- WS-23 Block (3): 0.5%: WS-23 block (3): 0.5%, no nicotine
- WS-23 Block (4): 1.0%: WS-23 block (4): 1.0%, no nicotine
- WS-23 Block (5): 2.0%: WS-23 block (5): 2.0%, no nicotine
- WS-23 Block (6): 4.0%: WS-23 block (6): 4.0%, no nicotine
Arm/Group | WS-3 Block (1): 0.05% | WS-3 Block (2): 0.1% | WS-3 Block (3): 0.5% | WS-3 Block (4): 1.0% | WS-3 Block (5): 2.0% | Menthol Block (1): 0.05% | Menthol Block (2): 0.1% | Menthol Block (3): 0.5% | Menthol Block (4): 1.0% | Menthol Block (5): 2.0% | WS-23 Block (1): 0.05% | WS-23 Block (2): 0.1% | WS-23 Block (3): 0.5% | WS-23 Block (4): 1.0% | WS-23 Block (5): 2.0% | WS-23 Block (6): 4.0%
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT05932693/Prot_SAP_000.pdf